CLINICAL TRIAL: NCT05539508
Title: Role of Peripheral Vision in Scene Perception
Brief Title: Role of Peripheral Vision in Scene Perception (PERISCE)
Acronym: PERISCE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01986-35
Record Dates: First submitted 2022-08-23; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Primary Open-angle Glaucoma (POAG)
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary open-angle glaucoma (POAG) group
  Interventions: Behavioral: Psychophysical evaluation
- Age-matched normally sighted control group
  Interventions: Behavioral: Psychophysical evaluation

INTERVENTIONS:
Behavioral: Psychophysical evaluation — All participants will be required to perform a short experiment on a computer (15 minutes) where they will look at different photographs of scenes of different luminance and spatial frequencies. They will have to perform various tasks on these images using the keys on the keyboard.

SUMMARY:
Despite its low spatial resolution, peripheral vision is very useful for rapidly categorizing a visual scene. Low spatial frequencies of a visual stimulus available in peripheral vision would allow a coarse categorization of the scene and objects (deciding, for example, whether it is an urban or natural landscape). This first representation would then trigger predictive mechanisms which would subsequently guide a more detailed visual analysis in central vision. The psychophysical studies that the investigators have already conducted in this scientific context has been carried out under normal vision conditions. The objective of this project is to study the influence of peripheral vision on central vision with an original approach: What are the consequences of a loss of peripheral vision on the processing performed in central vision? The project will concern patients with glaucoma. This ophthalmic pathology particularly affects the peripheral retina and thus represents a good pathological cognitive model of a visual recognition system in which peripheral vision is less important. The investigators will conduct psychophysical studies with glaucomatous patients and healthy volunteers with normal vision. All participants will be required to perform a short experiment on a computer (15 minutes) where they will look at different photographs of scenes of different luminance and spatial frequencies. Participants will have to perform various tasks on these images using the keys on the keyboard.

ELIGIBILITY:
Inclusion Criteria:

For patients :

* between 18 and 80 years old
* stable bilateral primary open angle glaucoma (POAG)
* visual acuity > 5/10 for distant vision for the eye tested
* peripheral visual field defect on the eye tested measured through a Humphrey Visual Field Analyzer

For healthy volunteers :

* between 18 and 80 years old
* visual acuity > 5/10
* absence of ophthalmologic disease other than Glaucoma (age-related macular degeneration, cataract except for uncomplicated cataract surgery, amblyopia, optic neuropathy, diabetic retinopathy …)

Exclusion Criteria:

* ophthalmologic disease other than Glaucoma (age-related macular degeneration, cataract except for uncomplicated cataract surgery, amblyopia, optic neuropathy, diabetic retinopathy …)
* treated with medication that might compromise sustained attention (benzodiazepine, narcoleptics)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: POAG patients and age-matched normally sighted controls
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Psychophysical measure : Percentage of correct response | Through study completion of 45 months
  Measure calculated by the comparison between the expected response and the response provided by the participant for each trial of the experiment
Psychophysical measure : Mean reaction time in milliseconds | Through study completion of 45 months
  Measure calculated by averaging the time in milliseconds taken by the participant to provide the response for each trial of the experiment

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be share in the context of publications through the Open Science Framework, a tool that promotes open, centralized workflows.
Time Frame: Data will become available after publications with no limit time
Access Criteria: Link to the Open Science Framework

REFERENCES:
- [Background] Roux-Sibilon A, Rutge F, Aptel F, Attye A, Guyader N, Boucart M, Chiquet C, Peyrin C. Scene and human face recognition in the central vision of patients with glaucoma. PLoS One. 2018 Feb 26;13(2):e0193465. doi: 10.1371/journal.pone.0193465. eCollection 2018. PMID 29481572
- [Background] Roux-Sibilon A, Trouilloud A, Kauffmann L, Guyader N, Mermillod M, Peyrin C. Influence of peripheral vision on object categorization in central vision. J Vis. 2019 Dec 2;19(14):7. doi: 10.1167/19.14.7. PMID 31826252
- [Background] Peyrin C, Roux-Sibilon A, Trouilloud A, Khazaz S, Joly M, Pichat C, Boucart M, Krainik A, Kauffmann L. Semantic and Physical Properties of Peripheral Vision Are Used for Scene Categorization in Central Vision. J Cogn Neurosci. 2021 Feb 11:1-15. doi: 10.1162/jocn_a_01689. Online ahead of print. PMID 33571079